CLINICAL TRIAL: NCT01959984
Title: Study on the Comparison Between"Standard Noodles" and Traditional Carbohydrates in the Diagnosis of Diabetes Mellitus.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, the vice-president of Shanghai Jiao Tong University Affiliated Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CCEMD018
Record Dates: First submitted 2013-09-29; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100g Standard Noodles (Experimental): 100g Standard Noodles
  Interventions: Other: 100g Standard Noodles
- 75g Oral Glucose (Experimental): 75g Oral Glucose
  Interventions: Other: 75g Oral Glucose

INTERVENTIONS:
Other: 100g Standard Noodles — Subjects are required to take 100g standard noodles,and then blood samples are collected at 0min,30min,60min,120min,180min.
  Arms: 100g Standard Noodles
Other: 75g Oral Glucose — Subjects are required to take 75g glucose solution,and then blood samples are collected at 0min,30min,60min,120min,180min.
  Arms: 75g Oral Glucose

SUMMARY:
The object of this study is to compare "100g Standard Noodles " with traditional carbohydrates including 75g glucose solution in 300ml water and 100g steamed bread in the diagnosis of diabetes mellitus.

In this study, we will compare the different effects of "100g Standard Noodles Tolerance Test"and "75g Oral Glucose Tolerance Test"on plasma glucose, insulin, c- peptide level and the relevant hormones level including glucagon-like peptide-1( GLP-1) and glucagon. Besides, in part of the subjects, the difference between "100g Steamed Bread Tolerance Test", "100g Standard Noodles Tolerance Test" and "75g Oral Glucose Tolerance Test" will be further evaluated.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

For healthy subjects:

1. Between 16-70 years old.
2. No weight fluctuation greater than 5% within 3 months.
3. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures .

For subjects with impaired glucose regulation(IGR):

1. Between 16-70 years old.
2. Impaired fasting glucose(IFG):6.1mM(109mg/ml)≤fasting plasma glucose(FPG)<7.0mM(126mg/ml),or impaired glucose tolerance(IGT):7.8mM（140mg/ml）≤2h plasma glucose(2hPG)<11.1mM(200mg/dl),or both.
3. No weight fluctuation greater than 5% within3 months.
4. Keep stable antidiabetic therapy for at least 2 months.
5. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures .

For subjects with type 2 diabetes mellitus(T2DM):

1. Between 16-70 years old.
2. T2DM:diabetic symptoms plus random blood glucose(RBG)≥11.1mM,or FPG ≥7.0mM(126mg/dl),or 2hPG ≥11.1mM(200mg/dl).
3. No weight fluctuation greater than 5% within 3 months.
4. Keep stable antidiabetic therapy at least for 2 months.
5. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.

For subjects with type 1 diabetes mellitus(T1DM):

1. Between 16-70 years old.
2. T1DM:diabetic symptoms plus RBG≥11.1mM,or FPG ≥7.0mM(126mg/dl),or 2hPG ≥11.1mM(200mg/dl).
3. Present at least one positive antibody of β cell including ICA,IAA,GADA,IA-2A and IA-2βA.
4. No weight fluctuation greater than 5% within 3 months.
5. Keep stable antidiabetic therapy for at least 2 months.
6. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.

Exclusion Criteria:

For healthy subjects:

1. Be diagnosed with diabetes or IGR in late 3 months.
2. With any significant medical condition,laboratory abnormality,or psychiatric disorders that will prevent the subject from participating in the study.
3. Any medical or surgical conditions possibly affecting the experiment result.
4. Participated in a clinical study involving administration of medication within 90 days.
5. Donated blood or plasma or had any other significant blood loss within 2 months.
6. Any clinically significant allergic diseases.
7. Recently drug or alcohol abuse(>35unit/week,1unit=8 g alcohol@1 standard drink@250ml beer@140ml wine@25ml strong alcohol drink like whiskey.)
8. Smokers or users of other tobacco products in the 3 months prior to screening.

For IGR and DM:

1. History of pancreatic diseases such as pancreatic cancer or pancreatitis.
2. Suffered from acute complications such as diabetic ketoacidosis and hyperosmolar coma within 3 months.
3. With any significant medical condition，laboratory abnormality,or psychiatric disorders that will prevent the subject from participating in the study.
4. Malignant tumor.
5. Being allergic to experiment arms.
6. Recently drug or alcohol abuse(>35unit/week,1unit=8 g alcohol@1 standard drink@250ml beer@140ml wine@25ml strong alcohol drink like whiskey.)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The plasma glucose level. | 12 months
  The primary outcome measures the plasma glucose level at 0min,30min,60min,120min,180min during "75g Oral Glucose Tolerance Test" and "100g Standard Noodles Tolerance Test" .
The insulin level. | 12 months
  The primary outcome measures the insulin level at 0min,30min,60min,120min,180min during "75g Oral Glucose Tolerance Test" and "100g Standard Noodles Tolerance Test" .
The c-peptide level. | 12 months
  The primary outcome measures the c-peptide level at 0min,30min,60min,120min,180min during "75g Oral Glucose Tolerance Test" and "100g Standard Noodles Tolerance Test" .

SECONDARY OUTCOMES:
The GLP-1 level. | 12months
  The outcome measures of the GLP-1 level at 0min,30min,60min,120min,180min during "75g Oral Glucose Tolerance Test" and "100g Standard Noodles Tolerance Test" .
The Glucagon level. | 12 months
  The outcome measures of the glucagon level at 0min,30min,60min,120min,180min during "75g Oral Glucose Tolerance Test" and "100g Standard Noodles Tolerance Test" .
The other relevant incretin hormones levels. | 12 months
  The outcome measures of the relevant incretin hormones level at 0min,30min,60min,120min,180min during "75g Oral Glucose Tolerance Test" and "100g Standard Noodles Tolerance Test" .
The plasma glucose, insulin, c-peptide and relevant incretin hormones level during "75g Oral Glucose Tolerance Test", "100g Standard Noodles Tolerance Test" and "100g Steamed Bread Tolerance Test". | 12 months

OTHER OUTCOMES:
Safety | 12 months
  Document the frequency and extent of side-effects.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD,PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ni M, Chen Y, Gu W, Zhang Y, Xu M, Gu Y, Chen Y, Zhu Y, Wang X, Luo Y, Xu Y, Lin X, Zeng YA, Liu R, Wang J. Association Between Circulating Gremlin 2 and beta-Cell Function Among Participants With Prediabetes and Type 2 Diabetes. J Diabetes. 2025 Apr;17(4):e70090. doi: 10.1111/1753-0407.70090. PMID 40270326